#### Subject information for the Polyethylene Wear Study on the Triathlon Knee Prosthesis

"Scientific research into the wear of two types of knee bearings"

Responsible researchers: Department: Orthopedics

Dear Sir / Madam,

As a follow-up to the conversation with your doctor, you will receive written information regarding a scientific study for which your cooperation has been requested.

We do not immediately ask you to make a decision. Please take a moment to reflect before you decide whether you want to participate or not. We recommend that you discuss your participation with your partner, family, doctor or others.

If you need to submit your questions to a doctor who is not directly involved in this study, you can find the name and telephone number of this independent doctor on the last page of this information letter.

#### 1. Purpose of the investigation

The purpose of the research for which we request your cooperation is to compare the anchoring and wear of two types of artificial knees. The best method to measure the artificial knee anchoring in the bone and the wear is with a so-called RSA (X-ray stereo photo grammetric analysis) photo. This is an X-ray with which the fixation of the artificial knee in the bone can be calculated. For this photo, a number of tantalum granules (Ø 1 mm) are inserted into the bone around the prosthesis during the operation.

#### 2. Which medical device is being investigated?

The orthopedics department of the Lange Land Hospital is conducting research into the functioning of knee prostheses. Total knee prostheses have been manufactured since 1993 and consist of an upper leg and lower leg component with the bearing in between: an intermediate piece of plastic (polyethylene). We look at the difference between two types of knee bearings. The one type of bearing, the N2Vac, is a widely used material with excellent wear prevention properties. The other type, X3, is a new generation to which even more durable properties are assigned.

#### 3. How is the investigation conducted?

If you decide to participate in this study, a draw will be used to determine the type of bearing you will receive. You have a 50% chance of getting the knee prosthesis with the N2vac lower, and a 50% chance of getting the knee prosthesis with the X3 lower. After the operation you will not be told which bearing you have received. The first RSA photo will be taken in the first week after your operation, after which you will be recalled at set intervals. Each visit, whether or not combined with the regular check-up and X-ray, will take approximately 20 minutes. During this visit you will be asked to complete 4 questionnaires that mainly deal with your health situation

#### 4. What is expected of you?

You must adhere to the rules of life that you are provided by your doctor and you must be present at all agreements made.

#### 5. What is more or different from the regular treatment you receive?

Regardless of whether you participate in this study or not, the medical treatment will be the same for both participants and non-participants in the first year after the operation, but there will be 1

additional check within the study. At every check-up, X-rays of your operated knee will be made, for participants also 1 extra photo will be made for the examination. If you participate in this study, you are also requested to participate in completing four questionnaires about your health and the knee prosthesis. It takes approximately 20 minutes to complete these questionnaires. You will receive the call for the outpatient checks at home. After 5 years the regular checks will take place again.

#### 6. What side effects can you expect?

This study does not expose you to risks other than the standard risks associated with total knee replacement surgery. Standard risks when placing a knee prosthesis include: anesthesia reactions, allergic reactions, risk of infection, damage to blood vessels and / or nerves, bone fracture or death. Your doctor will inform you sufficiently about this. The radiation load of the extra stake photos that are made is well within the range of radiation to which someone may be exposed each year.

#### 7. What are the possible pros and cons of participating in this study?

Although this research does not directly benefit you, we try to improve the results of this study, surgery techniques for placing knee prostheses, and the design of the knee prosthesis.

#### 8. What happens if I do not participate in the study?

If you decide not to participate in the study, it will not have any influence on the future level of care that you receive during treatment.

### 9. What happens if, after initially giving permission, you no longer wish to participate in this study?

Your participation in this research is voluntary. If you give permission to participate in this study, you have the freedom to reconsider that decision at any time. You do not have to give a reason for this, but you will be asked to do so out of interest. Your doctor may also stop your participation in the study if he or she believes that this is better in your situation. He or she will discuss this with you. If new information becomes known during the examination, your treating doctor will also discuss this with you. Whether or not to participate does not in any way affect your further treatment or the relationship with your doctor.

#### 10. What are the conditions for early termination of the study?

For medical reasons agreed upon by Stryker, the sponsor of this study and your responsible doctor, you may choose to discontinue the study. There are no risks associated with the premature termination of the study; you will simply continue to participate in the regular follow-up checks.

#### 11. Are you insured when you participate in the study?

The principal of this investigation has taken out insurance for the implementation of the investigation. More information about the insurance can be found in Appendix 2

### 12. Will you be informed if any relevant information about the study becomes known to you in the meantime?

You will be notified in writing of relevant information.

#### 13. What happens to your data?

All information about individual patients collected in the context of the study is only transmitted in coded form to the prosthetic producer and stored electronically for a maximum of 15 years. A separate legal description has been added for this in Appendix 1. In order to ensure that the investigation runs correctly, specialists and clinical investigation staff members directly

associated with this investigation may have access to your patient file and the report resulting from the investigation.

In addition, the national and foreign authorities responsible for clinical examinations, the Southwest Holland Medical Ethics Committee and employees of the knee prosthesis manufacturer are also authorized to see your patient's file and the report resulting from the examination from the doctor's investigator. However, they are required to maintain strict confidentiality and to comply with the Personal Data Protection Act. Data is also recorded in a computer file and on forms. By signing the consent form you give permission for this inspection, the recording of data. Your identity will also be treated confidentially when the research results are published. During your meeting with your doctor you will be informed orally and in writing about this study. A week before your surgery you will receive verbal information and the opportunity to ask questions, after which you also have a few days to change your mind. The investigator must be informed at least 2 days before the operation whether or not you are participating.

### 14. Is your doctor and / or treating specialist informed about participation?

Your doctor will not be informed about your participation in the study.

### 15. Are there any additional costs / reimbursement if you decide to participate in this study?

There are no additional costs, no expense allowance.

### 16. Which medical ethics review committee has approved this study?

METC Southwest Holland

#### 17. Do you want to know anything else?

If you have any questions regarding this investigation as a result of this information, you can contact your treating physician, the investigator or the independent physician, the latter is not directly involved in the investigation but is informed about the content. For general information about participation in scientific research, please refer to the brochure "Medical research". If you decide to participate in this research, we ask you to put a signature on the next page (the consent form). With the signing you indicate that you have received and understood this information and know what is expected of you with regard to the investigation. If there are any complaints, you can turn to the complaints officers of the 't Lange Land hospital: on behalf of Mrs. Z. Gerodimos - Smits or Mrs. J. Luitwieler-Bosma. They can be reached on telephone number: 079 - 346.24.16

#### 18. Attachments

- 1.Transfer of patient information
- 2. Insurance supplement
- 3. Medical scientific research

Kind regards,

Your treating physician 079-3462535 Independent doctor: Leiden University Medical Center 071-5263606

#### **Declaration of consent**

Polyethylene Wear Study on the Triathlon Knee Prostesis "Scientific research into two different types of knee bearings"

I have read the information letter for the test subject. I could ask additional questions. My questions have been answered enough. I had enough time to decide if I would like to participate.

I know that participating is completely voluntary. I know that I can decide at any time not to participate. I don't have to give a reason for that.

I know some people can see my data. Those people are listed in the General brochure.

I give permission to use my data for the purposes stated in the information letter. I give permission to keep data for a maximum of 15 years after the end of this study.

| I think it's good to participate in this study. |
|---|
| Surname and initials: |
| Signature: |
| Date: |
| The undersigned declares that the person mentioned above has been informed orally and in writing about the above-mentioned investigation. He / she also declares that a premature termination of participation by the above-mentioned person will have no influence whatsoever on the care that is due to him or her. |
| Name: |
| Position: |
| Signature: |
| Date: |

#### **ATTACHMENT 1**

This research involves the collection of data, possibly also personal data. This data can be kept by Stryker or subsidiaries of Stryker. By agreeing to the research, I authorize Stryker to transfer the data both internally (jointly owned with Stryker) and externally (third parties under contract) if this is done for scientific purposes. If data is transferred to a third party outside the EU / EEA, the receiving party must comply with the data protection laws of Switzerland, a country whose data protection laws are appropriate according to the European Commission and Stryker's headquarters are located in Europe. This permission can be withdrawn at any time, without impact on the appointment that your place arranges within the clinical investigation.

#### INFORMATION ABOUT THE INSURANCE

Everyone who participates in this study has an insurance policy. The insurance covers damage that is the result of participation in the study. This applies to damage that comes up during the investigation, or within four years after the end of the investigation. You must also have reported the damage to the insurer within those four years.

In the event of damage, you can go directly to the insurer or claims representative. The research insurer is:

Name: AON

Address: Paalbergweg 2-4

1105 AG Amsterdam

Telephone: 020-430 55 00

The claims adjuster of the investigation is:

Name: C.P.J. Verberne Address: Paalbergweg 2-4

1105 AG Amsterdam

Telephone: 020 430 5552

The insurance offers a maximum coverage of € 450,000 per test subject and € 3,500,000 for the entire study, and € 5,000,000 per year for all studies by the same client. The coverage of specific claims and costs is further limited to certain amounts. You will find this in the Decree on compulsory insurance for medical research involving people. Information about this can be found on the website of the Central Committee on Research related People: www.ccmo.nl.

A number of exclusions apply to this insurance. The insurance does not cover the following damage:

- Damage that, due to the nature of the investigation, was (almost) certain that it would occur;
- Damage to health that would also have occurred if you had not participated in the study;
- Damage that is the result of not (fully) complying with instructions or instructions;
- Damage to descendants, as a result of the adverse effect of the research on you or your offspring;
- For research into existing treatment methods: damage that is the result of one of these treatment methods:
- For research into the treatment of specific health problems: damage that is the result of non-improvement or deterioration of these health problems.

#### ATTACHMENT 1

This research involves the collection of data, possibly also personal data. This data can be kept by Stryker or subsidiaries of Stryker. By agreeing to the research, I authorize Stryker to transfer the data both internally (jointly owned with Stryker) and externally (third parties under contract) if this is done for scientific purposes. If data is transferred to a third party outside the EU / EEA, the receiving party must comply with the data protection laws of Switzerland, a country whose data protection laws are appropriate according to the European Commission and Stryker's headquarters are located in Europe. This permission can be withdrawn at any time, without impact on the appointment that your place arranges within the clinical investigation.

#### INFORMATION ABOUT THE INSURANCE

Everyone who participates in this study has an insurance policy. The insurance covers damage that is the result of participation in the study. This applies to damage that comes up during the investigation, or within four years after the end of the investigation. You must also have reported the damage to the insurer within those four years.

In the event of damage, you can go directly to the insurer or claims representative. The research insurer is:

Name: AON

Address: Paalbergweg 2-4

1105 AG Amsterdam

Telephone: 020-430 55 00

The claims adjuster of the investigation is:

Name: C.P.J. Verberne Address: Paalbergweg 2-4

1105 AG Amsterdam

Telephone: 020 430 5552

The insurance offers a maximum coverage of € 450,000 per test subject and € 3,500,000 for the entire study, and € 5,000,000 per year for all studies by the same client. The coverage of specific claims and costs is further limited to certain amounts. You will find this in the Decree on compulsory insurance for medical research involving people. Information about this can be found on the website of the Central Committee on Research related People: www.ccmo.nl.

A number of exclusions apply to this insurance. The insurance does not cover the following damage:

- Damage that, due to the nature of the investigation, was (almost) certain that it would occur;
- Damage to health that would also have occurred if you had not participated in the study;
- Damage that is the result of not (fully) complying with instructions or instructions;
- Damage to descendants, as a result of the adverse effect of the research on you or your offspring:
- For research into existing treatment methods: damage that is the result of one of these treatment methods;
- For research into the treatment of specific health problems: damage that is the result of non-improvement or deterioration of these health problems.

This is a non-certified translation of the patient informed consent and attachments as there was no requirement for an English version of a patient informed consent as the single center study occurred in the Netherlands. The original Dutch patient informed consent is as follows:

Proefpersoneninformatie ten behoeve van de Polyethylene Wear Study on the Triathlon Knee Prosthesis

"wetenschappelijk onderzoek naar de slijtage van twee soorten knielagers"

Verantwoordelijk onderzoekers: dhr. H.H. Kaptijn, dhr. R.de Ridder, dhr. P.T.H. Langendijk en

dhr. V.J. Rudolphy

Afdeling: Orthopaedie

Geachte mevrouw/ meneer,

In aansluiting op het gesprek met uw behandelend arts ontvangt u hierbij de schriftelijke

informatie met betrekking tot een wetenschappelijk onderzoek waarvoor uw medewerking is

gevraagd.

Wij vragen u niet onmiddellijk om een beslissing te nemen. Neemt u rustig enige bedenktijd

voordat u beslist of u meedoet of niet. Wij raden u aan om uw deelname te bespreken met uw

partner, familie, huisarts of anderen.

Mocht u behoefte hebben uw vragen voor te leggen aan een arts die niet direct bij dit onderzoek

betrokken is, dan kunt u de naam en het telefoonnummer van deze onafhankelijk arts vinden op

de laatste pagina van deze informatiebrief.

1. Doel van het onderzoek

Het doel van het onderzoek waarvoor wij uw medewerking vragen is om de verankering en

slijtage van twee typen kunstknieën te vergelijken. De beste methode om de kunstknie

verankering in het bot en de slijtage te meten is met een zogenaamde RSA (röntgen stereofoto

grammetrische analyse) foto. Dit is een röntgenfoto waarmee de fixatie van de kunstknie in het

bot berekend kan worden. Voor deze foto worden tijdens de operatie een aantal tantalium

korreltjes (ø 1mm) in het bot ingebracht rond de prothese.

2. Welk medisch hulpmiddel wordt onderzocht?

Op de afdeling orthopaedie van 't Lange Land Ziekenhuis wordt onderzoek verricht naar het

functioneren van knieprotheses. Totale knieprotheses worden sinds 1993 vervaardigd en

bestaan uit een bovenbeen en onderbeen component met daartussen de lager: een tussenstuk

van plastic (polyethyleen). Er wordt gekeken naar het verschil tussen twee typen knielagers. Het

Page 1 of 6

ene type lager, de N2Vac, is een veel gebruikt materiaal met uitstekende eigenschappen ter voorkoming van slijtage. Het andere type, X3, is een nieuwe generatie aan welke nog extra slijtvastere eigenschappen worden toegewezen.

#### 3. Hoe wordt het onderzoek uitgevoerd?

Als u besluit mee te werken aan dit onderzoek wordt door middel van loting bepaald welk type lager u krijgt. U heeft 50% kans op het krijgen van de knieprothese met de N2vac lager, en 50% kans op het krijgen van de knieprothese met de X3 lager. Na de operatie zal u niet verteld worden welke lager u heeft ontvangen. In de eerste week na uw operatie zal de eerste RSA foto gemaakt worden, waarna u op vaste intervallen opnieuw opgeroepen wordt. Elk bezoek, al dan niet gecombineerd met de reguliere controle en röntgenfoto, zal ongeveer 20 minuten in beslag nemen. Tijdens dit bezoek zal u gevraagd worden om 4 vragenlijsten in te vullen die voornamelijk gaan over uw gezondheidssituatie.

#### 4. Wat wordt er van u verwacht?

U dient zich te houden aan de leefregels die u, door uw behandelend arts, worden verstrekt en u dient bij alle gemaakte afspraken aanwezig te zijn.

#### 5. Wat is meer of anders dan de reguliere behandeling die u krijgt?

Ongeacht of u deelneemt aan dit onderzoek, of niet, de medische behandeling zal het eerste jaar na de operatie, voor zowel deelnemers als niet-deelnemers hetzelfde zijn, echter binnen de studie zal er nog 1 extra controle plaatsvinden.

Bij elke controle zullen er röntgenfoto's van uw geopereerde knie gemaakt worden, voor deelnemers wordt tevens ook 1 extra foto gemaakt ten behoeve van het onderzoek.

Indien u meedoet aan dit onderzoek wordt u ook verzocht om mee te werken aan het invullen van <u>vier vragenlijsten</u> over uw gezondheid en de knieprothese. Het invullen van deze vragenlijsten duurt ongeveer 20 minuten. De oproep voor de poliklinische controles ontvangt u thuis. Na 5 jaar zullen de gewone controles weer plaats vinden.

#### 6. Welke bijwerkingen kunt u verwachten?

U wordt met deze studie niet blootgesteld aan andere risico's dan de standaard risico's bij de totale knieprothese operatie. Standaard risico's bij het plaatsen van een knieprothese zijn bijvoorbeeld: reacties op de verdoving, allergische reacties, infectie gevaar, schade aan bloedvaten en/of zenuwen, breken van het bot of de dood. Uw arts zal u hier voldoende over

inlichten. De stralenbelasting van de extra rongenfoto's die gemaakt worden is ruim binnen de marge van straling waaraan iemand per jaar blootgesteld mag worden.

#### 7. Wat zijn de mogelijke voor-en nadelen van deelname aan dit onderzoek?

Hoewel u zelf niet direct baat heeft bij dit onderzoek, proberen we met de resultaten van dezestudie,operatietechnieken voor het plaatsen van knieprotheses, en het ontwerp van de knieprothese te verbeteren.

#### 8. Wat gebeurt er als ik niet deel neem aan de studie?

Als u besluit om niet deel te nemen aan de studie, zal dat geen enkele invloed hebben op de toekomstige mate van zorg die u ontvangt tijdens de behandeling.

U ontvangt de prothese, met N2Vac lager, zoals deze standaard wordt gebruikt in het ziekenhuis.

# 9. Wat gebeurt er als u, na in eerste instantie toestemming te hebben gegeven, niet meer wenst deel te nemen aan dit onderzoek?

Uw medewerking aan dit onderzoek is vrijwillig. Als u toestemming geeft om aan dit onderzoek mee te doen, heeft u te allen tijde de vrijheid om op die beslissing terug te komen. U hoeft hiervoor geen reden op te geven, wel wordt het u uit interesse gevraagd. Ook uw behandelend arts kan uw deelname aan het onderzoek stopzetten als hij of zij vindt dat dit in uw situatie beter is. Hij of zij bespreekt dat dan met u. Wanneer tijdens het onderzoek nieuwe informatie bekend wordt, zal uw behandelend arts dit eveneens met u bespreken.

Het wel of niet meedoen heeft op geen enkele wijze gevolgen voor uw verdere behandeling of de verstandhouding met uw arts.

#### 10. Wat zijn de voorwaarden voor voortijdig stopzetten van de studie?

Uit medische overwegingen overeengekomen door Stryker, de sponsor van deze studie en uw verantwoordelijk arts kan ervoor gekozen worden de studie stop te zetten.

Aan het voortijdig beeindigen van de studie zijn geen risico's verbonden, u zult weer gewoon deelnemen aan de reguliere na-controles.

#### 11. Bent u verzekerd wanneer u aan het onderzoek meedoet?

De opdrachtgever van dit onderzoek heeft voor de uitvoering van het onderzoek een verzekering afgesloten. Meer informatie over de verzekering kunt u vinden in bijlage 2

## 12. Wordt u geinformeerd als er tussentijds voor u relevante informatie over de studie bekend wordt?

U wordt schriftelijk op de hoogte gebracht van voor u relevante informatie.

#### 13. Wat gebeurt er met uw gegevens?

Alle in het kader van het onderzoek verzamelde gegevens over afzonderlijke patiënten worden uitsluitend in gecodeerde vorm schriftelijk doorgegeven aan de producent van de prothese en elektronisch maximaal 15 jaar opgeslagen. In bijlage 1 is hiervoor een aparte juridische beschrijving toegevoegd. Om een correct verloop van het onderzoek te waarborgen, mogen specialisten en klinisch onderzoek medewerkers direct verbonden aan dit onderzoek inzage krijgen in uw patientendossier en het uit het onderzoek resulterende rapport. Daarnaast zijn de voor klinische onderzoeken bevoegde binnen- en buitenlandse instanties, van de Medisch Ethische Commissie Zuidwest Hollanden medewerkers van de producent van de knieprothese ook bevoegd om bij de artsonderzoeker inzage te krijgen in uw patiëntendossier en het uit het onderzoek resulterende rapport. Zij zijn echter verplicht tot strikte vertrouwelijkheid en tot inachtneming van de wet bescherming persoonsgegevens. Er worden ook gegevens opgenomen in een computerbestand en op formulieren. Door ondertekening van het toestemmingsformulier geeft u toestemming voor deze inzage, de opname van gegevens.Uw identiteit wordt ook vertrouwelijk behandeld, wanneer de onderzoeksresultaten gepubliceerd worden. Tijdens uw gespek met uw arts zult u schriftelijk en mondeling worden geïnformeerd over deze studie. Een week voordat u geopereerd wordt krijgt u mondelinge informatie en de mogelijkheid om vragen te stellen, waarna u ook nog een paar dagen bedenktijd heeft. Minimaal 2 dagen voor de operatie moet de onderzoeker op de hoogte zijn of u wel of niet deelneemt.

# 14. Wordt uw huisarts enlof behandelend specialist geinformeerd bij deelname? Uw huisarts zal niet worden geinformeerd over uw deelname aan het onderzoek.

## 15. Zijn er extra kostenlis er een vergoeding wanneer u besluit aan dit onderzoek mee te doen?

Er zijn geen extra kosten aan verbonden, er wordt geen onkostenvergoeding betaald.

# 16. Welke medisch-ethische toetsingscommissie heeft dit onderzoek goedgekeurd? METC Zuidwest Holland

17. Wilt u verder nog iets weten?

Mocht u naar aanleiding van deze informatie nog vragen hebben met betrekking tot dit

onderzoek dan kunt u daarmee terecht bij uw behandelend arts, de onderzoeker of de

onafhankelijk arts, deze laatste is niet direct betrokken bij het onderzoek maar is wel inhoudelijk

op de hoogte. Voor algemene informatie over deelname aan wetenschappelijk onderzoek

verwijzen wij u naar de brochure " Medisch-wetenschappelijk onderzoek". Wanneer u besluit

aan dit onderzoek deel te nemen vragen we u op de volgende pagina (het

toestemmingsformulier) een handtekening te zetten. Met de ondertekening geeft u te kennen

dat u deze informatie ontvangen en begrepen heeft en weet wat er van u verwacht wordt met

betrekking tot het onderzoek.

Mochten er klachten zijn dan kunt u zich wenden tot de klachtenfunctionarissen van 't Lange

Land ziekenhuis: t.a.v. Mevrouw Z. Gerodimos – Smits of mevrouw J. Luitwieler-Bosma.

Zij zijn te bereiken op telefoonnummer: 079 – 346.24.16

18. Bijlagen

1. Overdracht patienteninformatie

2. Verzekeringsbijlage

3. Medisch-wetenschappelijk onderzoek

Met vriendelijke groet,

Uw behandelend arts

079-3462535

Onafhankelijk arts:

Prof.dr. R.G.H.H. Nelissen

Leids Universitair Medisch Centrum

071-5263606

#### **Toestemmingsverklaring**

#### Polyethylene Wear Study on the Triathlon Knee Prostesis

"Wetenschappelijk onderzoek naar twee verschillende typen knielagers"

Ik heb de informatiebrief voor de proefpersoon gelezen. Ik kon aanvullende vragen stellen. Mijn vragen zijn genoeg beantwoord. Ik had genoeg tijd om te beslissen of ik meedoe.

Ik weet dat meedoen helemaal vrijwillig is. Ik weet dat ik op ieder moment kan beslissen om toch niet mee te doen. Daarvoor hoef ik geen reden te geven.

Ik weet dat sommige mensen mijn gegevens kunnen zien. Die mensen staan vermeld in de Algemene brochure.

Ik geef toestemming om mijn gegevens te gebruiken voor de doelen die in de informatiebrief staan.

Ik geef toestemming om gegevens nog maximaal 15 jaar na afloop van dit onderzoek te bewaren. Ik vind het goed om aan dit onderzoek mee te doen.

| Achternaam en voorletters: |
|---|
| Handtekening: |
| Datum: |
| Ondergetekende verklaart dat de hierboven genoemde persoon zowel mondeling als schriftelijk over het bovenvermelde onderzoek is geïnformeerd. Hij/zij verklaart tevens dat een voortijdige beëindiging van de deelname door bovengenoemde persoon, van geen enkele invloed zal zijn op de zorg die hem of haar toekomt. |
| Naam: |
| Functie: |
| Handtekening: |
| Datum: |

#### **BIJLAGE 1**

Dit onderzoek houdt de inzameling van gegevens in, mogelijk ook van persoonsgegevens. Deze gegevens kunnen bijgehouden worden door Stryker of dochtervennootschappen van Stryker. Door in te stemmen met het onderzoek, geef ik Stryker mijn toestemming om de gegevens zowel intern (gemeenschappelijke eigendom met Stryker) als extern (derden onder contract) over te dragen indien dit gebeurt in het kader van wetenschappelijke doeleinden. Als er gegevens worden overgedragen aan een derde buiten de EU / EER, moet de ontvangende partij de gegevensbeschermingswetten naleven van Zwitserland, een land waarvan de gegevensbeschermingswetten volgens de Europese Commissie gepast zijn en Stryker's hoofkantoor van Europa is gevestigd. Deze toestemming kan te allen tijde ingetrokken worden, zonder impact op de afspraak die uw plaats binnen het klinisch onderzoek regelt.

#### INFORMATIE OVER DE VERZEKERING

Voor iedereen die meedoet aan dit onderzoek is een verzekering afgesloten. De verzekering dekt schade, die het gevolg is van deelname aan het onderzoek. Dit geldt voor schade die naar boven komt tijdens het onderzoek, of binnen vier jaar na het einde van het onderzoek. U moet de schade ook binnen die vier jaar aan de verzekeraar hebben gemeld.

In geval van schade kunt u zich direct wenden tot de verzekeraar of schaderegelaar.

De verzekeraar van het onderzoek is:

Naam: AON

Adres: Paalbergweg 2-4

1105 AG Amsterdam

Telefoonnummer: 020-430 55 00

De schaderegelaar van het onderzoek is: Naam: C.P.J. Verberne adres: Paalbergweg 2-4

1105 AG Amsterdam

Telefoonnummer: 020 430 5552

De verzekering biedt een maximumdekking van € 450.000 per proefpersoon en € 3.500.000 voor het gehele onderzoek, en € 5.000.000 per jaar voor alle onderzoeken van dezelfde opdrachtgever. De dekking van specifieke schades en kosten is verder tot bepaalde bedragen beperkt. Deze vindt u in het *Besluit verplichte verzekering bij medisch-wetenschappelijk onderzoek met mensen*. Informatie hierover kunt u vinden op de website van de Centrale Commissie Mensgebonden Onderzoek: www.ccmo.nl.

Voor deze verzekering gelden een aantal uitsluitingen. De verzekering dekt de volgende schade niet:

- schade waarvan op grond van de aard van het onderzoek (nagenoeg) zeker was dat deze zich zou voordoen;
- schade aan de gezondheid die ook zou zijn ontstaan als u niet aan het onderzoek had deelgenomen;
- schade die het gevolg is van het niet (volledig) nakomen van aanwijzingen of instructies;
- schade aan nakomelingen, als gevolg van een nadelige inwerking van het onderzoek op u of uw nakomeling;
- bij onderzoek naar bestaande behandelmethoden: schade die het gevolg is van één van deze behandelmethoden;
- bij onderzoek naar de behandeling van specifieke gezondheidsproblemen: schade die het gevolg is van uitblijvende verbetering of van verslechtering van deze gezondheidsproblemen.